CLINICAL TRIAL: NCT04050241
Title: Objective and Subjective Mental Workload During Direct and Indirect Laryngoscopy in Anesthetists: an In-vivo, Cross-over Randomized Study
Brief Title: Workload in Anesthesiological Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Principal Investigator, Eleonora Orena, Senior Researcher, Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: AR-INNCB-02-2011
Record Dates: First submitted 2019-08-01; First posted 2019-08-08 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Work Related Stress
Keywords: Mental workload; Anesthesia; Laryngoscopy; Intubation; Perceived workload
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videolaryngoscope (Experimental): Anesthetists performing intubation with the Glidescope videolaryngoscope.
  Interventions: Device: Glidescope intubation
- Direct laryngoscope (Experimental): Anesthetists performing intubation with the Mcintosh laryngoscope.
  Interventions: Device: Mcintosh intubation

INTERVENTIONS:
Device: Glidescope intubation — Anesthetists will perform intubation in patients undergoing elective neurosurgery with the Glidescope videolaryngoscope, while completing a secondary auditory task. Response times to the secondary task will be recorded, and operators will complete the NASA Task Load Index questionnaire at the end of each procedure.
  Arms: Videolaryngoscope
Device: Mcintosh intubation — Anesthetists will perform intubation in patients undergoing elective neurosurgery with the Mcintosh laryngoscope, while completing a secondary auditory task. Response times to the secondary task will be recorded, and operators will complete the NASA Task Load Index questionnaire at the end of each procedure.
  Arms: Direct laryngoscope

SUMMARY:
The study evaluates differences in perceived and objective workload in anesthetists during intubation procedure with a direct (Mcintosh) or indirect (Glidescope) laryngoscope. Expert anesthetists will perform 3 intubations per device, while completing a secondary task, during which reaction times to an auditory stimulus will be recorded, and will complete a questionnaire (the NASA-Task Load Index) to evaluate their perceived workload at the end of each procedure.

DETAILED DESCRIPTION:
Intubation and laryngoscopy are the most demanding procedure in anesthesiological routine clinical practice, associated with high workload. The measurement and management of workload is considered important in anesthesiology to prevent work-related stress and errors in performance. New devices, thanks to advances in technology, seem promising in reducing operators' workload and improving safety and success of intubation processes.

Therefore, in this study, based on previous results, the hypothesis that the Glidescope videolaryngoscope reduces operators' perceived and and objective workload, as compared to the standard Mcintosh laryngoscope, will be tested.

Expert anesthetists will perform 3 intubations per device in a randomized order, while completing a secondary task, during which reaction times (verbal responses) to an auditory stimulus (a clacson) will be recorded, and operators will complete a questionnaire (the NASA-Task Load Index) to evaluate their perceived workload at the end of each procedure.

ELIGIBILITY:
Inclusion Criteria:

* Anesthetists with expertise in videolaryngoscopy and direct laryngoscopy that give consent to participate

Exclusion Criteria:

* Anesthetists that refuse to participate
* Anesthetists without expertise in videolaryngoscopy and direct laryngoscopy that give consent to participate
* Anesthetists that have left hearing loss

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Perceived workload | Immediately after the procedure/intervention
  Results from the self-reported NASA Task Load Index will be considered as measure of perceived subjective workload

SECONDARY OUTCOMES:
Quantitative workload | During the laryngoscopy/intubation procedure
  Reaction times to a secondary auditory task will be used as a measure of mental workload

CONTACTS AND LOCATIONS:
Overall Officials: Elenora F Orena, PhD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy